CLINICAL TRIAL: NCT02290522
Title: A Prospective Study Using Genomic Screening to Select Patients for Targeted Molecular Treatment
Brief Title: Copenhagen Prospective Personalized Oncology (CoPPO)
Acronym: CoPPO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ulrik Lassen (Other)
Responsible Party: Sponsor-Investigator, Ulrik Lassen, MD, PH.D, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1300530
Record Dates: First submitted 2014-10-08; First posted 2014-11-14 (Estimated); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- tumor biopsy (Experimental): Tumor biopsy for targeted treatment according to molecular profile
  Interventions: Procedure: Tumor biopsy

INTERVENTIONS:
Procedure: Tumor biopsy — Biopsy of lesion for molecular characterization

SUMMARY:
Patients with advanced solid tumors referred to the Phase 1 Unit are offered mapping of GA for identification of pts who could benefit from a personalized treatment.

DETAILED DESCRIPTION:
Two ultrasound-guided biopsies obtained to be stored in RNAlater® for DNA and RNA purification. A 3rd biopsy for histology is paraffin embedded. SNP-array (Affymetrix Cytoscan HD) from DNA (tumor) is performed to identify copy number changes. Whole exome sequencing (WES) from DNA (tumor and blood) will be performed using sequence capture, SureSelect v5 (Agilent) and Illumina HiSeq2500 to call tumor specific mutations. Expression levels of therapeutic targets are revealed by expression Array from tumor RNA. In addition to the expression array, RNA-seq (Nugens Ovation RNA-seq system v2) is performed to investigate whether chromosomal translocations were the reason for tumor specific expression of an oncogene. Results will be reviewed by a tumor board. Patients with specific genetic profiles that can be targeted with marketed drugs or drugs under development are offered such treatment. PFS from the treatment is compared to PFS of the most recent standard treatment (PFS ratio).

ELIGIBILITY:
Inclusion Criteria:

* Solid tumor
* No standard treatment option
* PS 0-1
* Lesion assessable for biopsy
* Measurable disease
* Informed consent

Exclusion Criteria:

* Life expectancy < 3 months
* Bone marrow suppression
* Abnormal renal or hepatic function
* Serious concurrent medical conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2013-05; Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Median progression free survival (PFS) | Median time from date of randomization to date of progression or death, assessed up to 100 months
  From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months

CONTACTS AND LOCATIONS:
Overall Officials: Ulrik Lassen, MD, PH.D., Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

REFERENCES:
- [Derived] Jacobsen IC, Spanggaard I, Hojgaard M, Belcaid L, Qvortrup C, Yde CW, Schmidt AY, Nielsen FC, Willemoe GL, Dam MS, Lassen U, Staal Rohrberg K. Extensive genomic analysis in patients with KRAS-mutated solid tumors shows high frequencies of concurrent alterations and potential targets but has limited clinical impact. Acta Oncol. 2022 Dec;61(12):1499-1506. doi: 10.1080/0284186X.2022.2156809. Epub 2022 Dec 18. PMID 36529989
- [Derived] Tuxen IV, Rohrberg KS, Oestrup O, Ahlborn LB, Schmidt AY, Spanggaard I, Hasselby JP, Santoni-Rugiu E, Yde CW, Mau-Sorensen M, Nielsen FC, Lassen U. Copenhagen Prospective Personalized Oncology (CoPPO)-Clinical Utility of Using Molecular Profiling to Select Patients to Phase I Trials. Clin Cancer Res. 2019 Feb 15;25(4):1239-1247. doi: 10.1158/1078-0432.CCR-18-1780. Epub 2018 Oct 1. PMID 30274980